CLINICAL TRIAL: NCT00789217
Title: The Comparative Results of Penicillin Testing in Patients With History of Allergic Reactions to Betalactams Between Using In-house Penicillin Test Preparation and Commercial Available Penicillin Testing Kit
Brief Title: Penicillin Skin Testing in Patients With History of Allergic Reactions to Betalactams
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Jettanong Klaewsongkram, MD, Chulalongkorn University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Chula-ARC 001/08
Record Dates: First submitted 2008-11-07; First posted 2008-11-11 (Estimated); Last update posted 2010-11-29 (Estimated); Status verified 2010-11

CONDITIONS: Penicillin Allergy
Keywords: Penicillin; Beta-Lactams; Allergy; Hypersensitivity
MeSH Terms: conditions — Hypersensitivity | interventions — Intradermal Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- In-house penicillin testing preparation (Active Comparator): In-house penicillin testing prepared from alkali-treated penicillin G
  Interventions: Procedure: Immediate skin test
- Commercial penicillin test kit (Active Comparator): Commercial penicillin test kit order from Diater company
  Interventions: Procedure: Immediate skin test
- Penicillin G Sodium (Active Comparator): Penicillin G Sodium from routine clinical use
  Interventions: Procedure: Immediate skin test

INTERVENTIONS:
Procedure: Immediate skin test — Intradermal test with immediate reading
  Other Names: Intradermal test with reading at 15 minutes after injection

SUMMARY:
This study aims to compare the readings of skin testing results in patients with suspected penicillin allergy between in-house penicillin test preparation and commercial available penicillin testing kit.

DETAILED DESCRIPTION:
The results of skin test with immediate reading will be compared between alkali-treated penicillin G and DAP reagents from Diater

ELIGIBILITY:
Inclusion Criteria:

1. Patients with history of hypersensitivity reactions to betalactams; penicillin, aminopenicillins, and cephalosporins
2. 15-65 years of age

Exclusion Criteria:

1. On antihistamine/ cannot discontinue antihistamine before the test
2. Having asthma exacerbation
3. Being pregnant
4. Suffering from severe systemic disease/ in bad health

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-12; Primary Completion 2010-03 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The skin testing results of in-house penicillin skin test and Penicillin G Sodium compared to commercial penicillin testing kit | 1 year

SECONDARY OUTCOMES:
Clinical correlation and side effects | 1 year
Correlations between Penicillin skin test result with specific IgE and/or basophil activation test | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jettanong Klaewsongkram, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand

REFERENCES:
- [Derived] Wangrattanasopon P, Ruxrungtham K, Chantaphakul H, Buranapraditkun S, Klaewsongkram J. Alkali-treated penicillin G solution is a better option than penicillin G as an alternative source of minor determinants for penicillin skin test. Allergy Asthma Proc. 2012 Mar-Apr;33(2):152-9. doi: 10.2500/aap.2012.33.3496. PMID 22525392